CLINICAL TRIAL: NCT04834479
Title: Assessment of Accuracy of Ultrasonography in Diagnosis of Non-osseous Lateral Ankle Instability in Comparison With Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Raafat Fouad, MRFouad, Assiut University
Other Study IDs: 17100620
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Ultrasound Therapy; Complications
Keywords: Lateral ankle instability, US, MRI

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ankle US and Ankle MRI — Ankle US and Ankle MRI

SUMMARY:
Chronic ankle instability (CAI) is a condition that often develops after repeated ankle sprains, increasing the susceptibility of the ankle to move into excessive inversion when walking on unsteady surfaces. Approximately 74% of acute ankle sprains result in persistent symptoms, 30% of which progress to chronic ankle instability. Arthroscopic examination and magnetic resonance imaging (MRI) are considered the two most accurate methods of diagnosing injuries to lateral collateral ligaments. Ultrasound has been proven able to detect soft tissue injuries, However, the use of ultrasound and its' ability to accurately diagnose CAI is still under debate. The aim of this study is to investigate the diagnostic accuracy of ultrasonography for the assessment of non-osseous lateral ankle instability in comparison with magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is a condition that often develops after repeated ankle sprains, increasing the susceptibility of the ankle to move into excessive inversion when walking on unsteady surfaces. Approximately 74% of acute ankle sprains result in persistent symptoms, 30% of which progress to chronic ankle instability.[1-3] CAI is diagnosed in individuals who report pain and tenderness on the lateral aspect of the ankle, or persistent swelling and discomfort for greater than six months with a history of re-injury or clinical instability of the ankle joint.[4, 5] The primary cause of damage to the structural stability of the ankle joint is trauma by forced inversion and plantarflexion. The lateral collateral ligaments, which are more commonly affected by acute sprains, include the anterior talofibular ligament (ATFL), the calcaneofibular ligament (CFL), and the posterior talofibular ligament (PTFL). The ATFL is primarily responsible for preventing excessive supination and anterior translation, while also restricting plantar flexion and internal rotation.

Common diagnostic tools used to identify ankle instability include clinical testing (like Anterior Drawer Test), imaging and arthroscopy. Arthroscopic examination and magnetic resonance imaging (MRI) are considered the two most accurate methods of diagnosing injuries to lateral collateral ligaments. [7] In a retrospective study conducted by Joshy et al., in which 24 patients underwent arthroscopy and MRI of the ankle, MRI was found to have both high specificity (100%) and high sensitivity (100%) for ATFL disruption. [8-10] Ultrasound has been proven able to detect soft tissue injuries, and has even become the gold standard for the detection of injuries to the patellar and Achilles tendons. [2, 11] However, the use of ultrasound and its' ability to accurately diagnose CAI is still under debate.

When imaging the ankle, ultrasound should be able to detect synovial lesions, ligamentous injury, and distinguish soft tissue from osseous impingement.[8] Dynamic ultrasound should be also used to discover dislocation of the peroneal tendons, or intra-sheath dislocation, which is indicated by an intact retinaculum with subluxation of the peroneal tendons within the groove.[11] Aim of the work: The aim of this study is to investigate the diagnostic accuracy of ultrasonography for the assessment of non-osseous lateral ankle instability in comparison with magnetic resonance imaging (MRI).

Patients and Methods:

fifty four patients complaining of acute or chronic lateral ankle instability will be included in this study.

Inclusion criteria:

Patients complaining of acute or chronic lateral ankle instability.

Exclusion criteria:

* Previous ankle surgery
* Interventional intra-articular procedures (previous arthroscope, injections)
* Systemic inflammatory disorders (collagen diseases)
* Diagnosed osseous lesions.

Methods:

All patients will be subjected to:

Thorough history taking and clinical provisional diagnosis. Plain X-ray of the affected ankle in AP and lateral views to exclude any osseous lesions.

Real-time high resolution ultrasonography of the affected ankle joint MRI for the affected ankle joint.

Ultrasound Technique:

The ultrasonographic examination of the ankle begins with the patient in supine position. Longitudinal scanning of the ankle was first performed to get an overall view of the tibio-talar joint and to detect joint effusion. Thereafter, slight inversion of the foot is performed while the patient in the same position to examine the lateral collateral ligaments and peroneal tendons. The Anterior talo-fibular ligament (ATFL) is first examined in oblique transverse plane from the tip of lateral malleolus, antero-medially and slightly downward, till the talus. Then, the Calcaneo Fibular ligament (CFL) is examined in oblique longitudinal plane from the lateral malleolar tip downward and slightly backward to the lateral surface of the calcaneus.

Regarding the peroneal tendons, they are examined from their supra-malleolar musculo-tendinous junction, and then just behind the lateral malleolus till their infra-malleolar course in both longitudinal and transverse planes.

MRI examination All patients will have MRI imaging of the affected ankle(s) on a high field-strength scanners.

Positioning:

Every patient lies supine with the ankle and foot in neutral position and plantar flexion of 20-30 degrees for reducing the "magic angle" artifact. No movement allowed during examination by supporting the ankle using pads.

Protocol:

The patients are examined by different pulse sequences including T1, T2, proton density, gradient echo and STIR. The examinations will be done in different planes.

Our usual protocol of examination is Sagittal T1WIs, Axial T1WIs T2WIs and proton density images, coronal T1WIs as well as Sagittal or coronal STIR.

Other parameters applied include slice thickness ranged from 3 to 5 mm, matrix 256/192 or 512/224, number of excitation 2 to 3 and field of view ranged from 12 to 16 cm, better kept <14 cm.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of acute or chronic lateral ankle pain and instability.

Exclusion Criteria:

* Previous ankle surgery
* Interventional intra-articular procedures (previous arthroscope, injections)
* Systemic inflammatory disorders (collagen diseases)
* Diagnosed osseous lesion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: fifty four patients complaining of acute or chronic lateral ankle pain and instability will be included in this study.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2021-04-03 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
To study the accuracy, sensitivity and specificity of Ultrasonography in assessment of lateral ankle disorders causing ankle instability and pain in comparison to MRI. | 1 year
  To study the accuracy, sensitivity and specificity of Ultrasonography in assessment of lateral ankle disorders causing ankle instability and pain in comparison to MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Raafat, Study Chair — Assiut University
Locations (1):
- Mariana Raafat Fouad, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wikstrom EA, Hubbard-Turner T, McKeon PO. Understanding and treating lateral ankle sprains and their consequences: a constraints-based approach. Sports Med. 2013 Jun;43(6):385-93. doi: 10.1007/s40279-013-0043-z. PMID 23580392
- [Background] Radwan A, Bakowski J, Dew S, Greenwald B, Hyde E, Webber N. EFFECTIVENESS OF ULTRASONOGRAPHY IN DIAGNOSING CHRONIC LATERAL ANKLE INSTABILITY:A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2016 Apr;11(2):164-74. PMID 27104050
- [Background] Delahunt E, Bleakley CM, Bossard DS, Caulfield BM, Docherty CL, Doherty C, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Remus A, Verhagen E, Vicenzino BT, Wikstrom EA, Gribble PA. Clinical assessment of acute lateral ankle sprain injuries (ROAST): 2019 consensus statement and recommendations of the International Ankle Consortium. Br J Sports Med. 2018 Oct;52(20):1304-1310. doi: 10.1136/bjsports-2017-098885. Epub 2018 Jun 9. PMID 29886432
- [Background] Houston MN, Van Lunen BL, Hoch MC. Health-related quality of life in individuals with chronic ankle instability. J Athl Train. 2014 Nov-Dec;49(6):758-63. doi: 10.4085/1062-6050-49.3.54. PMID 25299444
- [Background] van Ochten JM, van Middelkoop M, Meuffels D, Bierma-Zeinstra SM. Chronic complaints after ankle sprains: a systematic review on effectiveness of treatments. J Orthop Sports Phys Ther. 2014 Nov;44(11):862-71, C1-23. doi: 10.2519/jospt.2014.5221. Epub 2014 Oct 9. PMID 25299494
- [Background] Croy T, Saliba SA, Saliba E, Anderson MW, Hertel J. Differences in lateral ankle laxity measured via stress ultrasonography in individuals with chronic ankle instability, ankle sprain copers, and healthy individuals. J Orthop Sports Phys Ther. 2012 Jul;42(7):593-600. doi: 10.2519/jospt.2012.3923. Epub 2012 Mar 23. PMID 22446334
- [Background] Polzer H, Kanz KG, Prall WC, Haasters F, Ockert B, Mutschler W, Grote S. Diagnosis and treatment of acute ankle injuries: development of an evidence-based algorithm. Orthop Rev (Pavia). 2012 Jan 2;4(1):e5. doi: 10.4081/or.2012.e5. Epub 2011 Dec 14. PMID 22577506
- [Background] Joshy S, Abdulkadir U, Chaganti S, Sullivan B, Hariharan K. Accuracy of MRI scan in the diagnosis of ligamentous and chondral pathology in the ankle. Foot Ankle Surg. 2010 Jun;16(2):78-80. doi: 10.1016/j.fas.2009.05.012. Epub 2009 Jul 8. PMID 20483139
- [Background] Jung HG, Kim NR, Kim TH, Eom JS, Lee DO. Magnetic Resonance Imaging and Stress Radiography in Chronic Lateral Ankle Instability. Foot Ankle Int. 2017 Jun;38(6):621-626. doi: 10.1177/1071100717693207. Epub 2017 Feb 1. PMID 28552041
- [Background] Morvan A, Klouche S, Thes A, Hardy P, Bauer T. Reliability and validity of preoperative MRI for surgical decision making in chronic lateral ankle instability. Eur J Orthop Surg Traumatol. 2018 May;28(4):713-719. doi: 10.1007/s00590-017-2116-4. Epub 2018 Jan 3. PMID 29299765